CLINICAL TRIAL: NCT02364167
Title: Acupuncture vs. Placebo Acupuncture and vs. Standard Therapy for Pain Control After Elective Caesarean Section - a Randomized Controlled Trial
Brief Title: Acupuncture for Pain Control After Elective Caesarean Section
Acronym: ACUSEC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC SC BB 04/15
Record Dates: First submitted 2015-02-09; First posted 2015-02-16 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Verum acupuncture (Experimental): Each patient will receive 16 permanent indwelling acupuncture needles, embedded in adhesive tape, bilaterally in addition to standard postoperative analgesia
  Interventions: Drug: Standard therapy; Device: Verum acupuncture
- Placebo acupuncture (Placebo Comparator): Each patient will receive 16 adhesive tapes mimicking the indwelling acupuncture needles bilaterally in addition to standard postoperative analgesia
  Interventions: Drug: Standard therapy; Other: Placebo acupuncture
- Standard therapy (Active Comparator): Each patient will receive just standard postoperative analgesia
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Standard therapy — Standard therapy includes pharmacologic treatment of postoperative pain according to the standards of our University hospital
  Other Names: Pharmacologic therapy of postoperative pain
Device: Verum acupuncture — Verum acupuncture will be performed using indwelling permanent acupuncture needles "New Pyonex" with 1,5 mm length, manufactured by Seirin Corp. Japan
  Arms: Verum acupuncture
Other: Placebo acupuncture — Placebo acupuncture will be performed using the placebo "New Pyonex" adhesive tapes, mimicking the needles, manufactured by Seirin Corp. Japan
  Other Names: Placebo
  Arms: Placebo acupuncture

SUMMARY:
The study entitled "Acupuncture vs. placebo acupuncture and vs. standard therapy for pain control after elective caesarian section - a randomized controlled trial" aims to investigate whether acupuncture with indwelling fixed needles reduces pain and analgesic requirement as compared to placebo and standard therapy in patients after after elective caesarian section (CS) in the period from January 2015 to May 2016.

For that purpose 180 adult patients scheduled to elective elective CS in spinal anesthesia will be recruited according to eligibility criteria. 120 patients will be randomized either to verum or placebo acupuncture, 60 patients will be included in non-randomized "standard therapy" arm. The outcome measures are: postoperative analgesic requirement, pain intensity, incidence of side effects and physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an American Society of Anaesthesiologists physical status of I to III scheduled for elective caesarean section in spinal anaesthesia
* Surgery time does not exceed 60 minutes
* Patients without previous opioid and psychotropic medication
* Patients ranged 19-45 years old
* Patients who have given written informed consent

Exclusion Criteria:

* Recidivist alcoholics
* Local skin infection at the sites of acupuncture
* Age < 19 and > 45 years
* Switching to general anaesthesia in cases where spinal anaesthesia fails
* Surgery time more than 60 minutes
* Intraoperative complications (bleeding, required blood transfusion more than 6 units of packed cells, cardiovascular instability, required catecholamines except for short hypotension after induction of spinal anaesthesia )
* Patients who consumed opioid medication at least 6 months before surgery
* Patients who are unable to understand the consent form and fill in the study questionnaire
* History of psychiatric disease

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Pain intensity as measured by Numeric Rating Scale 1-10 | 4:00 P.M. on the 1st postoperative day

SECONDARY OUTCOMES:
Total requirement of postoperative analgesics | 4:00 P.M. on the 2nd postoperative day
Incidence of complications and adverse effects | 4:00 P.M. on the 2nd postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Taras I Usichenko, MD, PhD, Study Director — University Medicine of Greifswald
Locations (1):
- Ernst Moritz Arndt University, Greifswald, Germany

REFERENCES:
- [Background] Usichenko TI. Acupuncture as part of multimodal analgesia after caesarean section. Acupunct Med. 2014 Jun;32(3):297-8. doi: 10.1136/acupmed-2014-010584. Epub 2014 May 7. No abstract available. PMID 24809368
- [Derived] Usichenko TI, Henkel BJ, Klausenitz C, Hesse T, Pierdant G, Cummings M, Hahnenkamp K. Effectiveness of Acupuncture for Pain Control After Cesarean Delivery: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e220517. doi: 10.1001/jamanetworkopen.2022.0517. PMID 35226080
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021